CLINICAL TRIAL: NCT04435288
Title: SPondyloArthritis: Inducing Drug-free Remission by Early TNF-Alpha bloCkade Under Guidance of Single Cell RNA Sequencing and Epigenetic Profiling. (The SPARTACUS Trial)
Brief Title: Spondyloarthritis: Inducing Drug-free Remission by Early TNF-alpha Blockade
Acronym: SPARTACUS
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BC-06226
Record Dates: First submitted 2020-06-09; First posted 2020-06-17 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Peripheral Spondyloarthritis

STUDY DESIGN:
Intervention Model Description: The SPARTACUS clinical trial consists of 2 phases (duration phase A is up to 60 weeks, phase B up to 3 years).
  SPARTACUS Phase A: "Remission-Induction Phase": (Baseline to (maximum) week 60) All patients (n=112) will be randomized (1:1) to either immediately receiving TNFi (golimumab) monotherapy ("TNFi Induction"-group) (n=56), or to the step-up regimen with csDMARDs ("csDMARD Step-up"-group) (n=56).
  SPARTACUS Phase B: "Drug-Free Remission Phase": cessation of therapy and exploration of drug-free remission in patients that achieve sustained clinical remission while on therapy in phase A (Duration: max. 3 years).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo controlled trial
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- TNFi-induction group (Active Comparator): The patients in the TNFi-induction group will receive golimumab at a standard dose of 50 mg subcutaneously (SC) every 4 weeks (with matching methotrexate (MTX)-placebo). In case of potential intolerance or toxicity to MTX-placebo, the dose will be gradually tapered to a minimum of 7.5 mg per week. When there are no tolerability/toxicity issues, the weekly dose of MTX-placebo will be increased to 20 mg at week 4. At week 12, a "Patient Acceptable Signs & Symptoms Improvement" ('PASSI') will be assessed by asking the question "Taking into account both efficacy and side effects, did you experience over the past 12 weeks enough improvement in signs and symptoms of your' arthritis-enthesitis-dactylitis to consider continuation of the same treatment schedule for the next 12 weeks?". If yes, all study medication will be kept stable until week 24; if no, oral sulphasalazine at a dose of 2 g per day will be started (escape medication).
  Interventions: Drug: week 24; Drug: week 36; Drug: Week 48; Drug: Week 60
- csDMARD-Step-up group (Active Comparator): The patients in the csDMARD-Step-up group will start with oral methotrexate (MTX) at a weekly dose of 15 mg for 4 weeks (with matching TNFi-placebo injections). In case of potential intolerance or toxicity to MTX , the dose will be gradually tapered to a minimum of 7.5 mg per week. When there are no tolerability/toxicity issues, the weekly dose of MTX will be increased to 20 mg at week 4. At week 12, a "Patient Acceptable Signs & Symptoms Improvement" ('PASSI') will be assessed by asking the question "Taking into account both efficacy and side effects, did you experience over the past 12 weeks enough improvement in signs and symptoms of your' arthritis-enthesitis-dactylitis to consider continuation of the same treatment schedule for the next 12 weeks?". If yes, all study medication will be kept stable until week 24; if no, oral sulphasalazine at a dose of 2 g per day will be started (escape medication).
  Interventions: Drug: week 24; Drug: week 36; Drug: Week 48; Drug: Week 60

INTERVENTIONS:
Drug: week 24 — At the week 24 timepoint, there are 3 possible scenario's:
  1. In patients that do not reach a state of clinical remission at week 24, blinded study medication will be interrupted and all patients will start open-label SC golimumab for an additional 36 weeks (up to max. week 60).
  2. In patients that achieve sustained clinical remission at week 24, defined as absence of clinical arthritis, enthesitis and dactylitis at both week 12 and week 24, all study medication will be discontinued and prospective follow-up will be planned in SPARTACUS Phase B.
  3. In patients that reach a state of clinical remission at week 24, but that did not yet reach this status at week 12, blinded study medication will be continued without any change in the treatment schedule for another 12 weeks.
Drug: week 36 — At week 36, patients that have continued the blinded study medication, will be re-assessed regarding sustained clinical remission (at week 24 and 36): if yes, all study medication will again be discontinued and prospective follow-up will be planned in SPARTACUS Phase B. If no, these patients will start open-label SC golimumab for an additional 24 weeks (up to max. week 60).
  If patients were in the "open-label golimumab treatment arm", effectiveness of the treatment will be assessed by using the "PASSI"-question. Inadequate responders will be discontinued from the study and will be treated with standard-of-care medication at the discretion of their treating rheumatologist, whereas patients with an acceptable improvement in signs and symptoms will continue with the same (open-label) medication schedule.
Drug: Week 48 — At week 48, all patients still remaining in SPARTACUS Phase A will have been treated with open-label golimumab (for a minimum of 12 weeks, but potentially up to 48 weeks). In patients reaching at this timepoint sustained clinical remission (at week 36 and 48), golimumab will be discontinued and prospective follow-up will be planned in SPARTACUS Phase B. For the other patients there are 3 possible scenarios:
  1. If clinical remission for the first time at week 48, continuation without any change in the treatment schedule for another 12 weeks.
  2. If an inadequate response (based on the "PASSI"-question), discontinuation from the study and standard-of-care medication
  3. If an acceptable improvement (but no clinical remission), continuation open-label golimumab for an additional 12 weeks, with open-label methotrexate (unless contra-indicated) to fulfil Belgian reimbursement criteria for TNFi.
Drug: Week 60 — At week 60 (final study visit of SPARTACUS Phase A), patients reaching sustained clinical remission (at week 48 and 60), will roll-over into SPARTACUS Phase B. All other patients will be discontinued and will be treated with standard-of-care medication (including TNFi, if in accordance with Belgian reimbursement criteria).

SUMMARY:
The SPARTACUS study will explore the therapeutic efficacy of 2 different treatment strategies for patients suffering from peripheral Spondyloarthritis (pSpA), classified according to the "Assessment in SpondyloArthritis international Society" (ASAS) classification criteria; it will be set up as a 48-week, prospective, randomized, active-comparator controlled, double-blind, double-dummy, clinical trial with a two-fold clinical objective:

* To compare a standard step-up approach using conventional synthetic Disease-Modifying Anti-Rheumatic Drugs (csDMARDs), such as methotrexate and/or sulphasalazine (the "csDMARD Step-Up"-strategy), with an early remission-induction treatment strategy that immediately introduces biological DMARDs (bDMARDs) as the first step in the treatment algorithm; in this group the Tumor Necrosis Factor inhibitor (TNFi) golimumab will be utilised (the "TNFi Induction"-strategy).
* To define the window of opportunity within which temporary treatment with bDMARDs might be more effective, by stratifying patients according to symptom duration: patients with shorter symptom duration (<3 months) versus those with more longstanding disease (between 3-12 months of symptom duration).

The double-blind phase of the study will compare the 2 treatment strategies with regard to the proportion of patients that achieve a status of (sustained) clinical remission. Differences between patients with very early disease (<3 months symptom duration) versus those with symptom duration between 3 and 12 months, will be evaluated.

In patients that reach sustained clinical remission, all study treatments (both in the "csDMARD Step-up"-group and the "TNFi Induction"-group) will be stopped, and long-term, clinical follow-up of these patients will allow to explore the possibility of "drug-free remission"; also with regard to this objective, the difference in symptom duration will be evaluated.

DETAILED DESCRIPTION:
SPARTACUS will have several achievable goals:

1. To show superiority of early treatment of pSpA patients with bDMARDs as compared to standard of care.

   In current practice, TNFi, the predominant bDMARDs in SpA, are only reimbursed in a restricted number of indications: they can be prescribed for axial disease (axSpA) and for the specific pSpA-entity, psoriatic arthritis (PsA); however, even in PsA, they are only reimbursed for longstanding, erosive disease, when patients have already failed (multiple) csDMARD(s). In patients with pSpA without psoriasis, rheumatologists can only prescribe csDMARDs, because TNFi are still off-label despite the overall good efficacy observed in several proof-of-concept studies, incl. one phase 3 trial (Ability-2). For this subgroup of patients, the unmet need is therefore still unacceptably high. Moreover, the patients included in Ability-2 reflected the current step-up treatment paradigm: patients already had longstanding disease (symptom duration of approx. 7 years) and had used (and failed) conventional treatment options before trial entry (99% prior use of Non-Steroidal Anti-Inflammatory Drugs (NSAIDs), 69% prior csDMARD use). In this population, a statistically significant difference between adalimumab and placebo was observed, but clinical remission rates remained somehow disappointing with only 33% of patients reaching the predefined remission outcome after 3 years of continuous adalimumab use.

   Until recently, no data were available regarding the treatment of early pSpA with bDMARDs. To address this knowledge gap, we designed a proof-of concept study to explore the therapeutic potential of TNFi in patients with pSpA with very short symptom duration, the CRESPA-trial. In this study, all patients had a symptom duration of less than 12 weeks: they were randomized to receive either immediate TNFi therapy (golimumab) or placebo. In summary, the results of this trial demonstrated that after 24 weeks of treatment, complete clinical remission could be achieved in 75% of golimumab-treated patients versus only 20% in patients treated with placebo (thus refuting the perception that a large majority of pSpA patients would go in spontaneous clinical remission). Due to the placebo-controlled design, the CRESPA trial did not provide any data on the percentage of patients that would have achieved clinical remission while on standard-of-care "csDMARD Step-up" treatment. The design of the SPARTACUS head-to-head trial will allow us to evaluate superiority of the new approach to current practice.
2. To delineate the window of opportunity for intensive treatment of pSpA: a transient time frame in which a disease is more susceptible to treatment.

   In the proof-of-concept CRESPA trial, all included patients had a symptom duration of less than 12 weeks. In these patients very high clinical remission rates were observed when patients were immediately treated with a TNFi. Interestingly, when the bDMARD treatment was interrupted after reaching sustained remission, 53% of patients remained in drug-free remission at long-term follow-up, providing preliminary evidence for the "window of opportunity" hypothesis: by effectively tackling pSpA (with bDMARDs) in a very early phase of the disease, drug-free remission might be an achievable goal in a significant number of patients. However, the CRESPA-trial does not allow to generalize the findings to pSpA patients with longer symptom duration. Moreover, the above-mentioned extension of the Ability-2 study would suggest that patients with a symptom duration of multiple years would have lower remission rates and would need chronic, life-long bDMARD treatment. The SPARTACUS trial will still focus on early treatment of pSpA (symptom duration <12 months), but the stratification of patients according to symptom duration (<3 months (identical to the CRESPA trial) versus between 3 and 12 months) will allow us to explore the exact time frame in which a window of opportunity is applicable. The goal is to demonstrate that drug-free remission is a feasible outcome when an early intensive treatment strategy is adopted and to delineate the window of opportunity (in terms of symptom duration) in which such a remission-induction strategy is successful, leading to significant health economic benefits.
3. To unravel new biomarkers of therapy response using cutting-edge single cell technology.

   In the CRESPA trial, we observed that despite the fact that 53% of patients were able to achieve drug-free remission, a significant proportion nevertheless relapsed. In this small proof-of-concept study, we were not able to detect significant predictors or remission or relapse. Also, 18% of patients did not achieve sustained clinical remission, but nevertheless experienced a significant improvement of signs and symptoms; in these patients long-term treatment was necessary. These results indicate that clinical response to TNFi is heterogeneous and underscores the need for biomarkers that can identify at baseline different pathogenic subsets that are associated with the (lack of) response to a TNFi. The recent introduction of new procedures such as ultrasound-guided synovial biopsy sampling in our early arthritis clinic has permitted to access synovial samples of virtually all peripheral joints (incl. wrists and small finger joints). By using innovative and unbiased tools recently developed in the area of single-cell analyses (RNA-sequencing and epigenetic profiling), we will obtain profound insights into the cellular heterogeneity of these unique patient samples.
4. To determine health-economic and societal impact of early, intensive bDMARD treatment of patients with recent-onset pSpA (compared to the currently reimbursed csDMARD Step-up strategy).

   A unique feature of SPARTACUS is that clinical trial and biomarker discovery will be coupled to calculation of the health-economic benefits of such an approach. We aim to determine from a healthcare and a societal perspective, the 2 years´ cost-utility, as well as a model-based lifelong incremental cost-utility of the innovative strategy compared to usual care. Uncertainty analyses will be performed and budget impact for the Belgian healthcare and social security (work disability) system will be calculated. Consistent with the increased call for transparency in health economic modelling, we aim to make our model available as a semi-open source model.
5. To increase awareness among referring physicians (general practitioners, other specialties that may evaluate patients with early SpA) and patient-advocacy groups about the value of early recognition and treatment in rheumatology.

It is still a great challenge to diagnose patients in an early stage of their disease. The delay between symptoms and diagnosis in SpA is still several years. As discussed above, it has been shown that in later stages of the disease, the treatment effect (even with bDMARDs) may be less impressive and chronic therapy is needed without possibility of drug withdrawal (leading to a high socioeconomic burden). The broad set-up of SPARTACUS across health institutes in Flanders will greatly facilitate the awareness and direct implementation of early arthritis strategies among physicians. Finally, results from SPARTACUS will provide evidence that will facilitate discussions with patients about treatment choices and ensure realistic treatment expectations and optimal health behaviour in patients with early pSpA.

ELIGIBILITY:
Inclusion Criteria:

SPARTACUS Phase A: "Remission-Induction Phase"

A subject will be eligible for study participation if all of the following criteria are met:

* Subjects must be able and willing to provide written informed consent and comply with the requirements of this study protocol.
* Subjects must be between 18 and 65 years of age.
* Subjects must have been diagnosed with peripheral spondyloarthritis by the treating rheumatologist.
* Subjects must meet the ASAS classification criteria for peripheral spondyloarthritis: subjects must have current arthritis (asymmetric or predominantly in the lower limbs) or current enthesitis (except for enthesitis only along the spine, sacroiliac joints and/or chest wall) or current dactylitis plus at least 1 of the following SpA features:

  * Anterior uveitis confirmed by an ophthalmologist (past or present)
  * Crohn's disease or ulcerative colitis diagnosed by a gastroenterologist (past or present).
  * Evidence of preceding infection (acute diarrhea or non-gonococcal urethritis or cervicitis 1 month before arthritis).
  * Psoriasis diagnosed by a dermatologist (past or present).
  * HLA B27 positivity
  * Sacroiliitis by imaging defined as bilateral grade 2-4 or unilateral grade 3-4 sacroiliitis on plain radiographs, according to the modified New York criteria or active sacroiliitis on MRI according to the ASAS consensus definition (ref of addendum).
* Subjects must have had onset of peripheral SpA symptoms ≤12 months prior to the screening visit.
* Subjects must have active disease at screening defined by Patient Global Assessment of Disease Activity Numerical Rating Scale (NRS) ≥ 4 and Patient Global Assessment of Pain NRS ≥ 4. At the baseline visit patients will be clinically evaluated to exclude spontaneous clinical remission.
* In subjects with concurrent axial SpA symptoms, the peripheral SpA symptoms must be the predominant symptoms at study entry based on the Investigator's clinical judgment.
* Subjects must have a negative PPD test (or equivalent) and chest radiography (anteroposterior and lateral view) at screening. If the subject has a positive PPD test (or equivalent), has had a past ulcerative reaction following PPD placement and/or a chest radiography consistent with prior TB exposure, the subject must initiate, or have documented completion of a course of anti-TB therapy.
* Women of childbearing potential or men capable of fathering children must be using adequate birth control measures during the study and for 3 months after receiving the last administration of study agent.
* Subject is judged to be in good health as determined by the principal investigator based upon the results of medical history, physical examination, laboratory profile, and chest x-ray (CXR) performed during screening.
* Subjects must be able and willing to self-administer SC injections or have a qualified person available to administer SC injections.

SPARTACUS Phase B: "Drug-Free Remission Phase"

A subject will be eligible for phase B of the study if all of the following criteria are met:

* Subjects must have participated in SPARTACUS Phase A.
* Subjects must have reached a status of sustained clinical remission (defined as absence of clinical arthritis, enthesitis and dactylitis at 2 consecutive 'major' visits with an interval of 12 weeks).

Exclusion Criteria:

* Medical history of inflammatory arthritis of a different etiology than peripheral spondyloarthritis (e.g. rheumatoid arthritis, systemic lupus erythematosus, gout, …).
* Prior adequate treatment with methotrexate and/or sulphasalazine.
* Prior exposure to any biologic therapy with a potential therapeutic impact on SpA.
* Treatment with any investigational drug of chemical or biological nature within a minimum of 30 days or 5 half-lives of the drug (whichever is longer) prior to the Baseline Visit.
* Subject is taking or has taken prohibited medications as outlined in Table 1 without meeting the mandatory washout period(s) relative to the baseline visit.
* Infection(s) requiring treatment with intravenous (iv) anti-infective agents within 30 days prior to the Baseline visit or oral anti-infectives within 14 days prior to the baseline Visit.
* Have a known hypersensitivity to human immunoglobulin proteins or other components of golimumab.
* History of central nervous system (CNS) demyelinating disease or neurologic symptoms suggestive of CNS demyelinating disease.
* History of listeriosis, histoplasmosis, chronic or active Hepatitis B infection, Hepatitis C infection, human immunodeficiency virus (HIV) infection, immunodeficiency syndrome, chronic recurring infections or active TB.
* (History of) chronic heart failure, including medically controlled, asymptomatic CHF.
* History of malignancy (including lymphoma and leukemia) other than a successfully treated non-metastatic cutaneous squamous cell or basal cell carcinoma or localized carcinoma in situ of the cervix.
* Have received any live virus or bacterial vaccination within 3 months prior to the first administration of study agent; patients who are expected to receive such vaccinations during the trial, or within 3 months after the last administration of study agent.
* Positive serum pregnancy test at screening.
* Female subjects who are breast-feeding.
* Clinically significant abnormal screening laboratory results as evaluated by the Investigator.
* Positive anti-cyclic citrullinated peptide (anti-CCP) antibody at screening if the titers are crossing 3 times the upper limit of normal.
* Subject is considered by the investigator, for any reason, to be an unsuitable candidate for the study.
* Subject with current symptoms of fibromyalgia that would confound evaluation of the patient.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical remission | 24 weeks
  At week 24 of the study the 2 treatment strategies will be compared with regard to achievement of clinical remission. Clinical remission is defined as complete absence of arthritis, dactylitis or enthesitis on clinical examination.

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Elewaut, Prof. dr, Principal Investigator — UZ Ghent; Filip Van den Bosch, Prof. dr, Principal Investigator — UZ Ghent; Philippe Carron, Dr., Principal Investigator — Uz Ghent
Locations (6):
- Belgium (6):
  - ASZ Aalst, Aalst
  - AZ Sint-Jan, Bruges
  - AZ Maria Middelares, Ghent
  - UZ Ghent, Ghent
  - UZ Leuven Gasthuisberg, Leuven
  - ZNA Jan Palfijn, Merksem

DOCUMENTS (1):
  • Study Protocol (2025-06-04): https://cdn.clinicaltrials.gov/large-docs/88/NCT04435288/Prot_000.pdf